CLINICAL TRIAL: NCT07324239
Title: Effect of TECAR Therapy on Pain and Quality of Life in Men With Chronic Prostatitis/Chronic Pelvic Pain Syndrome: a Randomized Controlled Trial
Brief Title: TECAR Therapy on Pain and Quality of Life in Men With Chronic Prostatitis/Chronic Pelvic Pain Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Middle East University (Other)
Responsible Party: Principal Investigator, Saher Lotfy El Gayar, Assistant Professor of Physical Therapy, Middle East University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TECAR therapy
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Prostatitis
MeSH Terms: conditions — Prostatitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TECAR therapy group (Active Comparator)
  Interventions: Device: TECAR therapy
- Control group (Sham Comparator)
  Interventions: Device: Sham TECAR therapy

INTERVENTIONS:
Device: TECAR therapy — WINBACK 3SE (France) will be used for TECAR therapy in this study. To facilitate optimal distribution of endogenous heat therapy and effective contact between the active electrodes, both capacitive and resistive, and the surface of the skin, a layer of high-conductivity cream will be applied to the treatment region. The plate, an inactive electrode, which has a specific size (21cm*15cm), will be placed on the gluteal region. The capacitive electrode was employed for a duration of seven and a half minutes, at an intensity of 30-40%, whereas the resistance electrode will be utilized for an equivalent period over the perineum at the same intensity.
  Arms: TECAR therapy group
Device: Sham TECAR therapy — The procedure is similar to the active treatment of TECAR, but with the critical difference being that the output intensity of the TECAR device will be set to zero during the session.
  Arms: Control group

SUMMARY:
Evaluate the effect of TECAR therapy on pain, voiding, erectile function, sleep quality and quality of life in men with chronic prostatitis/chronic pelvic pain syndrome.

DETAILED DESCRIPTION:
Sixty men with chronic prostatitis/chronic pelvic pain will be sourced from the urology outpatient clinic at Tanta University hospitals in Egypt, with referrals from urologists. Patients will be randomly assigned into two groups.

Study group: It will include 30 men receiving true TECAR therapy plus dietary and life style adjustments.

Control group: It will include 30 men receiving sham TECAR therapy plus dietary and life style adjustments.

Evaluation Procedures:

1. Pain, voiding, and quality of life using the National Institutes of Health-Chronic Prostatitis Symptom Index.
2. Sleep quality using the Pittsburgh Sleep Quality Index.
3. Erectile function using the International Index of Erectile Function.

ELIGIBILITY:
Inclusion Criteria:

* Presence of chronic prostatitis/chronic pelvic pain symptoms for more than 6 months.
* Ages will be ranged from 30 to 50 years old.

Exclusion Criteria:

1. Urinary and seminal infections.
2. Recent parenteral steroid administration.
3. Prior prostate or pelvic surgery.
4. Lower urinary tract disorders such as bladder stones.
5. Implanted electronic devices as pacemakers.
6. Sensory loss over the perineum.

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-07 (Estimated)

PRIMARY OUTCOMES:
Pelvic pain | Baseline and 8 weeks later
  Pain will be assessed using the National Institutes of Health-Chronic Prostatitis Symptom Index

SECONDARY OUTCOMES:
Quality of life of men | Baseline and after 8 weeks
  Quality of life will be assessed using the National Institutes of Health-Chronic Prostatitis Symptom Index

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Saif, Study Director — National institute for Gerontology
Locations (1):
- Tanta University Hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No